CLINICAL TRIAL: NCT00602732
Title: Intervention for Low-income Pregnant Women With Partner Abuse
Brief Title: Interpersonal Treatment Program to Prevent Depression and Post-Traumatic Stress Disorder in Low-Income Pregnant Women With Partner Abuse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH075013 (NIH); R34MH075013 (NIH); DSIR 83-ATP
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Depression, Postpartum; Depression
Keywords: Partner Abuse; Preventive Intervention; Postpartum Depression; Postpartum PTSD
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants assigned to the ROSE program
  Interventions: Behavioral: The Reach Out for a Safe Environment (ROSE) program
- 2 (Active Comparator): Participants assigned to enhanced care as usual
  Interventions: Behavioral: Enhanced care as usual (ECU)

INTERVENTIONS:
Behavioral: The Reach Out for a Safe Environment (ROSE) program — Participants in the ROSE program will receive a course on managing stress and negative feelings and will learn how to access resources for help. The ROSE program involves four 90-minute group sessions over a 4-week period prior to delivery. Participants will also attend one 50-minute booster session within 4 weeks prior to delivery of their babies.
  Other Names: Reach Out Stay Strong: Essentials for New Mothers
  Arms: 1
Behavioral: Enhanced care as usual (ECU) — Participants in ECU will receive the usual medical care provided for pregnant women at their prenatal clinic. Participants will also receive educational material and a list of treatment resources for depression.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of an interpersonally oriented treatment program called Reach Out for a Safe Environment in preventing depression and post-traumatic stress disorder in low-income pregnant women who have experienced recent partner abuse.

DETAILED DESCRIPTION:
Each year, approximately 324,000 pregnant women experience partner abuse (PA). With the emotional highs and lows that accompany new motherhood, pregnancy is often a challenging process for many women. Experiencing PA, while already going through a vulnerable time during pregnancy, may have harmful effects on the well-being of the woman and her infant. Women affected by PA are at an increased risk for certain physical and psychological problems, including depression and post-traumatic stress disorder (PTSD). Furthermore, the emotional distress from PA may impair a woman's ability to seek out the necessary support to ensure the safety of herself and her children. There have been few research efforts to develop an effective treatment to reduce the psychological impact of PA on pregnant women and even fewer efforts that target low-income women, who make up a large portion of affected women. The Reach Out for a Safe Environment (ROSE) program is an interpersonally oriented treatment developed to address factors that may contribute to postpartum mental health difficulties associated with PA. This study will evaluate the effectiveness of the ROSE program in preventing depression and PTSD in low-income pregnant women who have experienced recent PA.

Participation in this single-blind study will last approximately 29 weeks. All potential participants will answer an initial questionnaire concerning their history of physical, sexual, or emotional abuse in the past year. Selected participants will then undergo an interview about symptoms of depression, reactions to trauma, emotional difficulties, and alcohol and drug use. Participants invited to continue in the study will then be randomly assigned to the ROSE program or enhanced care as usual (ECU). Participants assigned to the ROSE program will attend four weekly 90-minute group sessions prior to delivery and one individual 50-minute booster session within 4 weeks of delivery. During these sessions, participants will learn ways to manage stress and negative feelings and how to access helpful resources. Participants will also complete two questionnaires about emotional difficulties per week for the duration of the program. Participants assigned to ECU will receive the usual medical care provided for pregnant women and will receive educational material on depression.

All participants will complete questionnaires and interviews about their emotional difficulties, relationships with others, and use of services for these difficulties prior to treatment assignment, 4 weeks after treatment assignment, 4 weeks after delivery, and 3 months after delivery. Participants in the ROSE program will additionally complete a questionnaire about their perceptions of the program after the fourth treatment session and after the booster session.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English sufficiently to complete the study procedures
* Willing and able to receive public assistance
* Identified as having experienced physical assault based on responses to CTS2 within 1 year prior to study entry
* 35 weeks or less gestation

Exclusion Criteria:

* Meets current criteria for major depressive disorder or post-traumatic stress disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-up Examination (LIFE) | Measured at Year 1

SECONDARY OUTCOMES:
Revised Conflict Tactic Scale (CTS2) | Measured at Year 1
Edinburgh Postnatal Depression Scale | Measured at Year 1
The Davidson Trauma Scale | Measured at Year 1
The Arizona Social Support Interview Schedule | Measured at Year 1
Parenting Stress Index | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Memorial Hospital, Providence, Rhode Island, United States